CLINICAL TRIAL: NCT01460251
Title: OPen Label Study to Evaluate Long Term Treatment Effect of DiaPep277 in Patients Who Have Completed Study 901 and Study 910 (Extension to 901 Phase III Study
Brief Title: OPen Label Study to Evaluate Long Term Treatment Effect of DiaPep277
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: rmc006492ctil
Record Dates: First submitted 2011-10-06; First posted 2011-10-26 (Estimated); Last update posted 2015-03-19 (Estimated); Status verified 2014-07

CONDITIONS: Type 1 Diabetes
Keywords: type 1 diabetes; beta cell; immunomodulation; immunointervention
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Drug:Diapep277 (Experimental): 1.0 mg DiaPep277® administered every 3 months.For patients who just completed the 2-year 901 study, a 3-year extended treatment will be offered with 13 administrations; patients who completed the 2-year 910 extension study will be offered a 3rd year of treatment with 5 additional administrations.
  Interventions: Drug: DiaPep277

INTERVENTIONS:
Drug: DiaPep277 — 1.0 mg DiaPep277® administered every 3 months.For patients who just completed the 2-year 901 study, a 3-year extended treatment will be offered with 13 administrations; patients who completed the 2-year 910 extension study will be offered a 3rd year of treatment with 5 additional administrations.

SUMMARY:
The study is an open-label extension study, offering patients who participated and completed previous studies 901 and 910 (an extension to 901) to continue treatment with DiaPep277 and clinical follow-up, for up to 3 additional years.The aim of the study is to collect safety and efficacy data of long term treatment effect of Diapep277.Only patients who completed studies 901 or 910 and still have stimulated C-peptide level equal to or above 0.2 nmol/L will be eligible for this extension study

DETAILED DESCRIPTION:
The study is an open-label extension study, offering patients who participated and completed previous studies 901 and 910 (an extension to 901) to continue treatment with DiaPep277 and clinical follow-up, for up to 2 additional years.The aim of the study is to collect safety and efficacy data of long term treatment effect of Diapep277.Only patients who completed studies 901 or 910 and still have stimulated C-peptide level equal to or above 0.2 nmol/L will be eligible for this extension study. The optimal dose and dosing regimen for this study will be the same as applied in the phase 3 study (901) and its extension study protocol (910), namely 1.0 mg DiaPep277® administered every 3 months. These conditions were determined as optimal based on the outcome of the phase 2 studies. For patients who just completed the 2-year 901 study, a 3-year extended treatment will be offered with 13 administrations; patients who completed the 2-year 910 extension study will be offered a 3rd year of treatment with 5 additional administrations.

ELIGIBILITY:
Inclusion Criteria:

* A patient that participated in Study 901 and received all doses of study medication, per protocol or Study 910 and received all doses of study medication, per protocol.
* Evidence of clinically significant residual beta-cell function demonstrated by MMTT stimulated C-peptide concentrations ≥ 0.20 nmol/L.
* If a female is of childbearing potential, the subject is not pregnant or lactating, and will use oral hormonal contraception or other equally effective contraceptive methods throughout the study.
* Stable medical condition for diseases, other than diabetes, during 30 days before the Screening Ext Visit.
* Signed informed consent to participate in the study
* The subject is on intensive insulin therapy (basis / bolus insulin) or is willing to initiate intensive insulin therapy, or is using an insulin pump. Patients on conventional insulin regime that had HbA1c<7% over the last 6 months can be recruited without switching to intensive insulin regime.

Exclusion Criteria:

* The subject has any significant diseases or conditions, including psychiatric disorders and substance abuse that, in the opinion of the Investigator, are likely to affect the subject's response to treatment or the ability to complete the study.
* The subject has a history of any kind of malignant tumor (not including basal cell skin cancer).
* The subject has clinical evidence of any diabetes-related complication that in the opinion of the Investigator would interfere with the subject's participation in and/or completion of the study.
* Subject has history of endogenous allergic reactivity
* The subject has known allergy to lipid emulsions.
* The subject has a known immune deficiency from any disease, or a condition associated with an immune deficiency.
* The subject is receiving immunosuppressive or immunomodulating agents or cytotoxic therapy or any medication that in the opinion of the Investigator might interfere with the study.
* The subject has any of the following clinically significant laboratory abnormalities:Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) greater than three times the upper limit of the normal (ULN) at the Screening-Ext Visit.Total bilirubin greater than 1.3 times the ULN at the Screening-Ext Visit.Subjects with severe renal failure at the Screening-Ext visit Clinically significant laboratory abnormalities, confirmed by repeat measurement,which may interfere with the assessment of safety and / or efficacy of the study drug, other than hyperglycemia and glycosuria at the Screening- Ext Visit.Fasting triglycerides >1000 mg/dL (11.3 mmol/L) at the Screening-Ext Visit. Suitable medical therapy for treatment of hyperlipidemia is allowed.
* The subject is a known or suspected drug abuser.
* The subject is known to test positive for HIV antibodies.
* The subject has chronic hematologic disease.
* The subject has liver disease such as cirrhosis or chronic active hepatitis.
* The subject has received any investigational drug within 3 months prior to Visit 12, other than DiaPep277 that was administered during study 901 or 910.
* The subject has had a severe blood loss within 2 months before the first dose of the study medication.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2012-01; Primary Completion 2014-12 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Adverse events | month 38
DiaPep277-specific antibodies | month 38

SECONDARY OUTCOMES:
Beta cell function-AUC of stimulated C-peptide from stimulated MMTT measured by radioimmunoassay | month 38
Percentage of patients that maintain stimulated C-peptide >/= 0.2nmol/L | month 38
percentage of patients that achieve glycemic target of HbA1c</=7% | month 38
Daily insulin dose adjusted to body weight at study end | month 38

CONTACTS AND LOCATIONS:
Overall Officials: Liat de Vries, Dr, Principal Investigator — Rabin Medical Center
Locations (2):
- Israel (2):
  - Hadassah Medical Center, Jerusalem
  - Schneider Children's Medical Center, Petah Tikva